CLINICAL TRIAL: NCT01653405
Title: Improving Anticoagulation Control in VISN 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDP 12-249
Record Dates: First submitted 2012-07-06; First posted 2012-07-31 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-01

CONDITIONS: Anticoagulants; Atrial Fibrillation; Venous Thromboembolism
Keywords: anticoagulants; pharmacists; quality improvement; quality of health care
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): VA patients treated at anticoagulation clinics at 8 sites in VISN 1. The intervention included a system to measure processes of care relevant to warfarin management, along with targeted audit and feedback.
  Interventions: Other: Multifaceted behavioral intervention
- Control Group (No Intervention): VA patients treated at anticoagulation clinics at 116 sites outside of VISN 1.

INTERVENTIONS:
Other: Multifaceted behavioral intervention — The intervention included access to a system to measure processes of care relevant to warfarin management, along with targeted audit and feedback.
  Arms: Intervention Group

SUMMARY:
Over 100,000 VHA patients receive anticoagulants (blood thinners) each year to prevent blood clots (including strokes). Too much anticoagulation increases the risk of serious or even fatal bleeding, and too little anticoagulation fails to protect the patient against blood clots. VHA anticoagulation clinics vary widely on how much time their patients spend in the therapeutic range, the range within which they are protected from clots but not at excessive risk of bleeding. Anticoagulation clinics can improve anticoagulation control by following several relatively simple procedures, including following-up promptly when patients are out of range and focusing on educating and supporting patients with poor control. In this study, the investigators will promote these practices at the anticoagulation clinics of the New England VA region, with a goal of improving anticoagulation control.

DETAILED DESCRIPTION:
Background: Over 100,000 VA patients receive oral anticoagulation (AC) each year to prevent blood clots, including strokes. AC is safer and more effective when it is managed skillfully and therefore well-controlled. AC control can be measured using percent time in therapeutic range (TTR), the proportion of time when patients are sufficiently anticoagulated to prevent clots but not excessively anticoagulated (which increases the risk of bleeding). The investigators have shown that the anticoagulation clinics (ACCs) of the VA vary widely on TTR, from 40% (very poor control) to 70% (excellent control). Improving TTR in the VA would prevent thousands of adverse events, including strokes, major hemorrhages, and deaths. The investigators have further investigated the structures and processes of care that contribute to these wide disparities in TTR performance.

Objectives: We applied proven methods to change provider behavior. The goal was to facilitate the adoption of these evidence-based practices in order to improve TTR in VISN 1. We utilized educational outreach, audit and feedback, internal facilitation, and external facilitation to promote improvements in three evidence-based processes of care; namely, follow-up within 7 days after deranged INR values, minimizing loss to follow-up, and use of guideline concordant INR targets.

Methods: Our clinician-focused intervention used a Dashboard to measure site-level TTR and processes of care and an Algorithm for routine AC management. Both the Dashboard and the Algorithm are concrete representations of our main evidence-based recommendations to improve AC management. We promoted their use through quarterly visits to the sites, at which we delivered audit and feedback and educational outreach, and also provided external facilitation to address ways to improve these performance measures. Our main outcome was change in site TTR over time, which was compared between VISN 1 and non-VISN 1 sites using an interrupted time series. Secondary outcomes included site-level changes in processes of anticoagulation care (measured using automated data). We used a difference-in-differences (DID) model to examine changes in anticoagulation control, measured as percent time in target range (TTR), as well as process measures, and compared VISN 1 sites to 116 VA sites located outside VISN 1. The pre-intervention period was from 5/1/10-5/1/13, while the post-intervention period was from 5/2/13-5/10/16.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving long-term oral anticoagulation with warfarin within the VA New England Region ("VISN 1")

Exclusion Criteria:

* Patients with valvular heart disease, who may have an INR target range other than 2-3. This usually represents between 10-15% of patients receiving anticoagulation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260576 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Borzecki, MD MPH, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rose AJ, McCullough MB. A Practical Guide to Using the Positive Deviance Method in Health Services Research. Health Serv Res. 2017 Jun;52(3):1207-1222. doi: 10.1111/1475-6773.12524. Epub 2016 Jun 28. PMID 27349472
- [Result] Rose AJ, Park A, Gillespie C, Van Deusen Lukas C, Ozonoff A, Petrakis BA, Reisman JI, Borzecki AM, Benedict AJ, Lukesh WN, Schmoke TJ, Jones EA, Morreale AP, Ourth HL, Schlosser JE, Mayo-Smith MF, Allen AL, Witt DM, Helfrich CD, McCullough MB. Results of a Regional Effort to Improve Warfarin Management. Ann Pharmacother. 2017 May;51(5):373-379. doi: 10.1177/1060028016681030. Epub 2016 Dec 17. PMID 28367699

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: VA sites
Groups:
- VISN1 (Intervention Group): VA patients receiving care at anticoagulation clinics at 8 sites within VISN 1
- Outside VISN1 (Control Group): VA patients receiving care at anticoagulation clinics at 116 sites outside of VISN 1.
Period: Overall Study
Arm/Group | VISN1 (Intervention Group) | Outside VISN1 (Control Group)
Started | 11794; 8 VA sites | 1248782; 116 VA sites
Completed | 8029; 8 VA sites (These patients had enough data to calculate TTR.) | 179979; 116 VA sites (These patients had enough data to calculate TTR.)
Not Completed | 3765; 0 VA sites | 1068803; 0 VA sites

BASELINE CHARACTERISTICS:
Population: Analysis was conducted at the site level and not the patient level.
Groups:
- Intervention Group: VA patients receiving anticoagulation clinic services at 8 sites in VISN 1.
- Control Group: VA patients receiving anticoagulation clinic services at 116 sites outside of VISN 1.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 8029 | 179979 | 188008
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (11.0) | 75.3 (11.2) | 75.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 4340 | 4521
  Male | 7848 | 175639 | 183487
Average TTR [Mean (Standard Deviation); unit: percentage of time in target INR range] | 66.4 (3.4) | 65.9 (3.7) | 65.9 (3.7)
Percentage of instances where INR<=1.5 was followed by a second INR within 7 days [Number; unit: percentage of instances] — Participants can contribute more than one instance each.
  percentage of instances | 36 | 28 | 28
Percentage of instances where an INR >= 4.0 was followed by a second INR within 7 days [Number; unit: percentage of instances] — Participants can contribute more than one instance each.
  percentage of instances | 50 | 42 | 42
Gaps in monitoring per patient-year [Mean (Standard Deviation); unit: gaps per patient-year] — Mean gaps in monitoring per patient year of therapy
  gaps per patient-year | 0.31 (0.15) | 0.37 (0.18) | 0.37 (0.18)
Percentage of patients whose mean INR value was between 2.3 and 2.7 [Number; unit: percentage of patients] | 50 | 47 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Time in Therapeutic Range (TTR)
Description: We compared TTR after the intervention to before the intervention. We used a difference in differences analysis to compare the absolute percentage change over time in the intervention group vs. the control group.
Time Frame: Baseline and 4 years
Population: Patients receiving care at specified sites. Patient-level analyses were aggregated to the site level.
Measure: Number; unit: percent change
Groups:
- Intervention Group: VA patients receiving anticoagulation clinic services at 8 sites within VISN 1. We provided sites with a system to measure processes of care, along with targeted audit and feedback. We focused on processes of care associated with site level anticoagulation control, including prompt follow-up after out-of-range international normalized ratio (INR) values, minimizing loss to follow-up, and use of guideline-concordant INR target ranges.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 8029 | 179979
percent change | 2.8 | 0.5
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p < 0.001, Difference in differences

2. Secondary Outcome: Change in Gaps in Monitoring Per Patient-year Among Patients Receiving Anticoagulation With Warfarin
Description: We compared the rate of 56-day gaps per patient year in the pre-intervention and post-intervention period. We used a difference in differences analysis to compare the intervention and control group. We are reporting absolute change.
Time Frame: Baseline and 4 years
Measure: Mean (Standard Deviation); unit: gaps per patient year
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 8029 | 179979
gaps per patient year | -0.03 (0.10) | -0.01 (0.09)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.43, test of differences

3. Secondary Outcome: Change in Percentage of Patients With Follow-up Within 7 Days After a High INR Value (>4.0)
Description: We compared the percentage of patients with follow-up within 7 days before and after the intervention. We used a difference in differences analysis to compare the intervention and control groups.
Time Frame: Baseline and 4 years
Measure: Number; unit: percentage change
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 8029 | 179979
percentage change | 15 | 0
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p < 0.001, difference in differences

4. Secondary Outcome: Change in Percentage of Patients With Follow-up Within 7 Days After a Low INR Value (1.5 or Lower)
Description: We compared the percentage of patients before and after the intervention. We used a difference in differences analysis to compare the intervention and control groups. Absolute percentage is reported.
Time Frame: Baseline and 4 years
Measure: Number; unit: percentage change
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 8029 | 179979
percentage change | 15 | 2
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p < 0.001, Difference in differences

5. Secondary Outcome: Percentage of Patients With Mean INR Value Between 2.3 - 2.7
Description: We compared the absolute percentage of patients with a mean INR of 2.3 - 2.7 before and after the intervention. We used a difference in differences analysis to compare the intervention and control groups.
Time Frame: Baseline and 4 years
Measure: Number; unit: percentage change
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 8029 | 179979
percentage change | 6 | 1
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.002, difference in differences

ADVERSE EVENTS:
Description: Adverse events were not monitored or assessed.
Arm/Group | VISN1 (Intervention Group) | Outside VISN1 (Control Group)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes